CLINICAL TRIAL: NCT03430557
Title: To Evaluate the Efficacy of Platelet Rich Plasma(PRP) in the Healing of Through and Through Periapical Lesions.
Brief Title: Platelet Rich Plasma in Healing of Through and Through Periradicular Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ritika
Record Dates: First submitted 2018-02-06; First posted 2018-02-13 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Periapical Lesions
Keywords: Endodontic surgery

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Periapical surgery with PRP (Experimental): MTA Retrograde filling will be performed after apicectomy for involved teeth and PRP will be filled in the lesion before closure of flap
  Interventions: Procedure: PRP
- Periapical surgery without PRP (Active Comparator): MTA Retrograde filling will be performed after apicectomy for involved teeth and flap will be closed without placement of PRP
  Interventions: Procedure: periapical surgery without PRP

INTERVENTIONS:
Procedure: PRP — platelet rich plasma
  Arms: Periapical surgery with PRP
Procedure: periapical surgery without PRP — retrograde MTA filling will be done after apicectomy and flap will be closed without filling anything in the bony lesion.
  Arms: Periapical surgery without PRP

SUMMARY:
Title : Evaluation of the efficacy of Platelet Rich Plasma (PRP) in healing of through and through lesions

Rationale: Bone replacement analogues have been used in the healing after periapical surgery. It has been a controversial issue to use bone grafts due to varied outcomes of different studies showing both improved outcomes and no difference. Lacunae while using bone grafts is their radiopacity which compounds the radiographic incomplete or uncertain healing. Thence we will be using platelet rich plasma as bone filling material.

Aims and Objectives : To evaluate outcome of platelet rich plasma in healing after periapical surgery for through an through lesions.

Setting: Department of Conservative Dentistry and Endodontics, PGIDS, Rohtak, Haryana.

Study Design: Randomized controlled trial

Time frame: 12-18 months

Population/participant : Patients of age 16-45 years (male/female) will be enrolled in the study with diagnosis of through and through lesions.

Inclusion criteria:- Patients of age 16 -45 years, -ve response to sensibility test, failed previous rct with purulent discharge, recurrent episode of purulent discharge.

Exclusion Criteria:- Unrestorable tooth, fractured /perforated roots, serious medical illness, smokers, pregnant females and lactating mothers, grade 3 mobile teeth, the need for antibiotic prophylaxis prior to dental care.

Sample size - a sample size of 30 patients has been calculated with n=15 in each group.

Methods- Clinically and radiographically diagnosis of lesion, sensibility test by heat, cold, EPT, preoperative evaluation by bleeding on probing, clinical attachment level, gingival marginal position & pocket depth. Surgical procedures will be carried out under operating microscope with 8 × 16 magnification by following standardized treatment methods.

Outcome Measures- The primary outcome variables observed for the study will be 3,6,9,12 months clinical and radiographic success rates in terms of resolution of periapical radiolucency using the same criteria as preoperatively on the radiograph and alleviation of clinical sign and symptoms.

Statistical Analysis : Intergroup and intra group comparison will be done according to distribution of data. Categorical data will be analyzed using chi-square test. Regression analysis will be done to observe any association between dependent and independent variables.

DETAILED DESCRIPTION:
The research process will be carried out in the Department Of Conservative Dentistry and Endodontics, Post Graduate Institute of Dental Sciences, Rohtak. Patients with through and through periradicular lesions diagnosed radiographically and clinically will be included in the study.

INCLUSION CRITERIA :-

1. Patients of age 16-45 years with a clinical & radiographic diagnosis of through and through periradicular lesion through CBCT.
2. Negative response to sensibility tests with radiographic evidence of periapical radiolucencies.
3. Failed previous root canal treatment with purulent discharge and radiographic evidence of periapical pathology.
4. Recurrent episode of purulent discharge and adequate final restoration with no clinical evidence of coronal leakage.

EXCLUSION CRITERIA :-

1. Unrestorable tooth
2. Fractured /perforated roots
3. Serious medical illness (uncontrolled/poorly controlled diabetes, unstable or life Threatening conditions or requiring antibiotic prophylaxis)
4. Smokers
5. Pregnant females and lactating mothers
6. Grade 3 mobile teeth

BASELINE PARAMETERS:

Endodontic evaluation - Pulp sensibility testing will be performed with a combination of heat test , cold test and electric pulp test. Teeth not responding to both thermal and electric test will be considered non vital.

Radiographic evaluation - Radiographs with paralleling cone technique will be taken at baseline and at subsequent appointments at standardized exposure parameters.

Clinical Periodontal Evaluation - The following clinical parameters will be evaluated at baseline and at subsequent follow up appointments in the test tooth and the contra lateral normal tooth in the same patient

1. Bleeding on probing - The presence or absence of bleeding following pocket probing will be recorded at 6 sites per tooth - mesiobuccal, buccal, distobuccal, mesiolingual, midlingual, distolingual.
2. Probing pocket depth (PPD) - Probing depth will be measured as the distance from the gingival margin to the base of the clinical pocket. The probing depth measurements will be assessed using a calibrated manual periodontal Williams 0 probe. The probe will be inserted with a firm, gentle pressure to the bottom of the pocket and maintained parallel to the vertical axis of the tooth. Measurements will be noted at 6 sites per tooth- mesiobuccal, midbuccal, distobuccal, mesiolingual, midlingual, distolingual. Measurements will be rounded to the nearest whole millimeter.
3. Clinical Attachment Level (CAL) - Clinical Attachment Level will be measured as the distance between the base of the clinical pocket and a fixed point on the crown, the cementoenamel junction (CEJ). Measurements will be made at 6 sites per tooth- mesiobuccal, midbuccal, distobuccal, mesiolingual, midlingual, distolingual using wiliiams 0 probe. Measurements will be rounded to the nearest whole millimeter. The mean CAL over all examined surfaces will be calculated.
4. Gingival marginal level/position from CEJ will be measured.

SAMPLE SIZE DETERMINATION:

A total of 30 patients (n=15 in each group) will be included in the study. A power calculation that was based on the previous data of different studies suggested ta sample size with 15 patients in each group.

RANDOMIZATION Patients will be randomly allocated by envelope method into two groups. Group I=PRP group, group II=Control group (CG).

SURGICAL TECHNIQUE :

With the exception of incisions, flap elevation and suturing, all surgical procedures will be performed under operating microscope in an operating room under 8x to 16x magnification.

The full thickness (mucoperiosteal flap) will be reflected under aseptic condition by technique-

1. Preoperative mouth rinse with 0.2% chlorhexidine mouthwash will be used.
2. Local anaesthesia with lidocaine 2% with epinephrine 1:80,000 will be achieved.
3. Buccal intrasulcular incision will be given up to the alveolar crest including one tooth mesial to the lesion & one tooth distal to the lesion, using no.15 blade on handle.
4. Mesial and distal vertical releasing incision will be given.
5. Full thickness flap will be gently reflected towards the apical area by periosteal elevator. The flap will be frequently irrigated with sterile saline to prevent dehydration of periosteal surface.
6. After complete elevation of the flap, debridement (periradicular curettage -enucleation) of the bony lesion will be performed. For additional hemostasis during surgery, cotton pellets soaked in 0.1% epinephrine will be applied topically as required.
7. A 2-3mm root tip with a 0º to 10º bevel angle will be sectioned with cylindrical surgical carbide burs at high speed with sterile water coolant.
8. Root end preparations extending 3mm into the canal space along the long axis of the root will be made by using a piezoelectric ultrasonic system with double angled Retrotips coated with Diamond abrasives.
9. Isthmuses, fins, and other significant anatomic irregularities will be identified in high magnification and will be treated with the ultrasonic instruments. Then the resected root surfaces will be stained with methylene blue and will be inspected with micromirrors under high magnification of 24x to examine the cleanliness of the root end preparation and detect any other overlooked anatomic details.
10. Root end filling will be done with mineral trioxide aggregrate (MTA). The adaptation of the filling material to the canal apical walls will be confirmed with the aid of an operating microscope at high magnification.
11. In control group cases wound site will be closed and sutured with 4-0 silk suture after irrigating the defect properly.
12. In test group cases PRP preparation will be performed by procedure described by okuda et al and hirmath et al. before surgery 8.5 ml blood will be drawn by venipuncture of anticubital vein and will be collected in 10 ml sterile glass tube coated with anticoagulant.
13. Whole blood will be centrifuged (2400rpm for 10 mins) to separate PRP and platelet poor plasma. PRP and PPP will be centrifuged again to separate PRP from PPP.
14. Fifteen minutes before use of the PRP , the PRP will be rapidly thawed, and a coagulated preparation of 0.3 mL of PRP will be obtained by its activation. Within a few minutes, the PRP preparation assumed a sticky gel consistency.

    Then PRP will be carried and packed into the defect to the level of defect walls .
15. Wound will then be closed and sutured the same way as control group.

PLATELET RICH PLASMA

Platelet Rich Plasma (PRP) is the component of blood in which the platelets are concentrated in a limited volume of plasma .This autologous plasma is a rich source of growth factors and its application is thought to be an effective way of inducing tissue repair and regeneration.

Numerous studies have shown PRP to be effective at promoting regeneration in both endodontic and periodontal defects.

It was also speculated that, because of its fibrinogen content, PRP reacts with thrombin and induces fibrin clot formation, which, in turn, is capable of upregulating collagen synthesis in the extracellular matrix and provides a favorable scaffold for cellular migration and adhesion.

POSTOPERATIVE INSTRUCTIONS:

The patients will be advised to avoid mouth rinsing, hard and hot food, hot drinks, heavy physical work, and tooth brushing during the day of surgery. Ice packs will be provided after surgery (10-20 minutes every 1 hour for a total of 3 applications).

POSTOPERATIVE FOLLOW UP:

Clinical and radiographic examinations will be performed every 3, 6 and 12 months by assessing the same parameters as baseline except that PD will not measured until 12 months. Routine examination procedure will be used to evaluate any evidence of signs and/or symptoms.

Radiographs will be taken at 3, 6 and 12th month of follow up. Radiographic healing will be assessed by the criteria :

1. Complete healing
2. Incomplete healing
3. Uncertain healing
4. Unsatisfactory healing

PROCESSING OF DATA

Inter and intra observation of data will be analyzed by distribution of data. Categorical data will be analyzed by chi square test. Regression analysis will be done to observe any association between independent and dependent variables. Interobserver/intraobserver reliability with cohen kappa analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of age 16-45 years with a clinical & radiographic diagnosis of through and through periradicular lesion through CBCT.
2. Negative response to sensibility tests with radiographic evidence of periapical radiolucencies.
3. Failed previous root canal treatment with purulent discharge and radiographic evidence of periapical pathology.
4. Recurrent episode of purulent discharge and adequate final restoration with no clinical evidence of coronal leakage.

Exclusion Criteria:

1. Unrestorable tooth 2. Fractured /perforated roots 3. Serious medical illness (uncontrolled/poorly controlled diabetes, unstable or life Threatening conditions or requiring antibiotic prophylaxis) 4. Smokers 5. Pregnant females and lactating mothers 6. Grade 3 mobile teeth

-

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
CHANGE IN PERIAPICAL RADIOLUCENCY ON RADIOGRAPH | Baseline to 1 year
  Radiographs will be taken at an interval of every 3 months for 1 year with the help of CDR DICOM. The lesion will be categorised as complete healing,incomplete healing,uncertain healing and failure.
  cllinical and radiographic examination will be performed at 3,6,9 and 12 months on same parameters as baseline except PD,CAL and GMP will not be measured till 12 months

SECONDARY OUTCOMES:
Clinical attachment level | Baseline to 1 year
  at the end of 1 year clinical attachment level will be checked for involved teeth.
Probing depth | Baseline to 1 year
  probing depth of the involved teeth will be checked at the end of 1 year.

IPD SHARING:
Plan to Share IPD: No